CLINICAL TRIAL: NCT00158379
Title: Carboplatin With Following Taxol® Therapy Under Additional Application of Epoetin Alfa (ERYPO ®) With Female Patients With Advanced Ovarian Cancer FIGO IA/G3 - IV
Brief Title: Taxol Carboplatin and Erythropoetin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3002000
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — 4 cycles of Carboplatin AUC 5 every 3 weeks. 12 weekly infusions of 80 mg/m² Taxol®

SUMMARY:
Time to progression (physical examination and radiologic imaging

ELIGIBILITY:
Inclusion Criteria:

* patients with primary ovarian cancer
* ECOG- 0-2
* Age >= 18
* no chemotherapy, radiation or immunotherapy in medical history for ovarian cancer
* adequate bone marrow, liver and kidney reserve: leukocytes ≥ 2.0 x 109/l, platelets ≥ 100 x 109/l, bilirubin <= 2,0 mg%, creatinine <= 1,5 mg% or creatinine clearance ≥ 60 ml/ min, hemoglobin ≥ 9 g/ dl SGOT, SGPT an AP within 3 fold of the reference laboratory's normal range
* written informed consent

Exclusion Criteria:

* before-existing heart illness, Cardiac infarct within last 6 months
* Radiotherapy within 4 weeks for study entry
* Patients in pregnancy or breast feeding (in premenopausal women anticonception has to be assured: intrauterine devices, surgical methods of sterilization, or, in hormone insensitive tumors only, oral, subcutaneous or transvaginal hormonal, non-estrogen containing contraceptives)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2003-07; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli, Principal Investigator — Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.noggo.de

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: July 2003 - December 2004
Period: Overall Study
Arm/Group | Paclitaxel
Started | 105
Completed | 105
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel
Number analyzed (Participants) | 105
Age, Continuous [Median (Full Range); unit: years] | 60.4 [23.4 to 80.3]
Gender [Count of Participants; unit: Participants]
  Female | 105
  Male | 0
Region of Enrollment [Number; unit: participants]
  Germany | 105

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival. Progression is Defined According WHO-criteria as Appearance of Any New Lesion or Increase of Existing Lesions by at Least 25%
Description: Time to progression
Time Frame: every 3 months for up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel
Number analyzed (Participants) | 105
months | 28.8 [25.4 to 40.0]

2. Secondary Outcome: Toxicity
Description: defined as hematological and non-hematological adverse events of grade >= grade 1
Time Frame: after every cycle during therapy phase and after every 3 months during follow-up, for up to 3 years
Measure: Number; unit: participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 105
participants | 105

ADVERSE EVENTS:
Arm/Group | Paclitaxel
Serious Adverse Events (participants affected / at risk) | 13/105
Other Adverse Events (participants affected / at risk) | 105/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel (N=105)
Nausea (Gastrointestinal disorders) | 2 (3)
Death (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Suspected thrombosis (Vascular disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 3 (3)
deterioration of general condition (General disorders) | 5 (5)
embolism (Vascular disorders) | 2 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel (N=105)
Anemia (Blood and lymphatic system disorders) | 105 (178)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No